CLINICAL TRIAL: NCT05430165
Title: Using Data-Adaptive Methods to Optimize Follow Up Of Injured Patients After Hospital Discharge in Cameroon (Aim 1)
Brief Title: Trauma Follow-Up Prediction (Project 2: Aim 1)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mefire Alain Chichom (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); University of California, Los Angeles (Other); University of California, Berkeley (Other)
Responsible Party: Sponsor-Investigator, Mefire Alain Chichom, Professor of Surgery, University of Buea
Organization: University of Buea (Other)
Other Study IDs: GRANT13254336; U54TW012087 (NIH)
Record Dates: First submitted 2022-06-05; First posted 2022-06-24 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Trauma; Injury Traumatic; Injuries
Keywords: Cameroon; Sub-Sahara Africa; mHealth
MeSH Terms: conditions — Wounds and Injuries | interventions — Triage; Equipment and Supplies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aim 1 Prospective Cohort: All eligible admitted trauma patients in the trauma registry and a qualitative study of 110 in-depth interviews (IDIs).
  Interventions: Other: Standard mHealth screening (triage) tool

INTERVENTIONS:
Other: Standard mHealth screening (triage) tool — Standard mHealth triage tool administered to eligible trauma patients by phone at 2 weeks, 1 month, 3 months, and 6 months post-hospital discharge. The mHealth triage tool is a survey that includes a 7-item questionnaire to identify their need for follow-up care.
  The need for follow-up care at any of the 4 follow-ups is defined as a flagged response to ≥1 question on the 7-item screening survey.

SUMMARY:
Traumatic injury and inadequate follow-up care are a significant cause of morbidity and 10% of all deaths in sub-Saharan Africa (SSA). In Cameroon, ~50% of all emergency department (ED) visits are due to traumatic injury, which is likely only ~60% of all traumatic injuries. In the subset of patients who seek care, follow-up after discharge can save lives, yet is uncommon due to both supply-side (e.g., under-resourced health systems, poor data) and demand-side (e.g., poverty) barriers, resulting in preventable complications after discharge (e.g., sepsis, osteomyelitis). Consequently, better follow-up care of trauma patients is a neglected, but high-yield opportunity to improve injury outcomes, especially when coupled with mobile health technologies (mHealth) to better predict and implement post-discharge care, preventing disability and death.

Thus, in this study, the investigators will scale up an existing trauma registry and expand use of a mHealth screening tool (triage tool). At 10 hospitals, the investigators will implement a trauma registry and mHealth tool and evaluate success in a mixed-methods study; a quantitative prospective cohort of all eligible injured patients will be followed for 6 months after discharge and an inductive qualitative study.

DETAILED DESCRIPTION:
Injury is the largest contributor to the global burden of surgical disease and the cause of 10% of all deaths in Sub-Saharan Africa (SSA). In SSA countries like Cameroon, injured people face multiple obstacles to trauma care, including potentially lifesaving follow-up care after hospital discharge. To significantly improve health in the SSA, there is an urgent need for effective, innovative, and scalable approaches to reduce morbidity and mortality from injury. Follow-up care of trauma patients is a neglected, but high-yield opportunity to improve injury outcomes, especially when coupled with mobile health technologies (mHealth) to better predict and implement post-discharge care. The ubiquity and high penetration of mobile phones in Cameroon provides a novel opportunity to improve injury care in the country. The long-term goal of this project is to improve trauma outcomes and reduce the burden associated with injury in Cameroon, with the overall objective of preventing disability and death.

A critical barrier to improved trauma outcomes in resource-limited SSA contexts is the rapid identification of patients who would benefit from further care and successful retention of these patients through treatment completion. Building on the investigators established research infrastructure in Cameroon, using an implementation science approach, the team will conduct a mixed-methods study and first expand the existing trauma registry to 10 hospitals and scale-up an mHealth, phone-based screening tool (triage tool) to identify trauma patients in Cameroon who would benefit from further formal medical care post-discharge. The second part of the study will consist of an inductive qualitative study using in-depth interviews (IDIs) with all the stakeholders: patients, ED staff, and CTR and mHealth research staff. In addition to the IDIs, the research team will also conduct a non-participant observation of the project's implementation, analyzing the behaviors of each stakeholder and the dynamics of interactions between them. The project's implementation will be assessed using domains of the Consolidated Framework for Implementation Research (CFIR) as theoretical framework. These data gathered in this aim will be triangulated to guide adaptation and optimization of the intervention in Aim 2.

ELIGIBILITY:
Inclusion Criteria:

Trauma Registry (CTR): Patients satisfying the following inclusion criteria will be included in the registry:

1. Patients with acute traumatic injury i.e. within 2 weeks of presentation for care.
2. Trauma patients who are formally admitted to the hospital as in-patients.
3. Trauma patients who die upon arriving to the Emergency Departments or while admitted in the hospital.
4. Trauma patients who are transferred to other health facilities.
5. Trauma patients with indications for hospital admission (based on physicians' assessments) but leave against medical advice
6. Trauma patients who are kept under observation in the Emergency Department for over 24 hours

Standard mHealth Triage Tool Eligibility: The mHealth triage tool will be administered to the subset of patients included in the trauma registry who are admitted then discharged home after treatment.

Exclusion Criteria:

Trauma Registry Exclusion criteria: Patients will not be excluded based on age, gender, race, or nationality. If patients or their surrogate decision-maker do not give consent to participation, those patients will be excluded.

According to the World Health Organization (WHO) injury definition, the following will be excluded from the definition of "injury": "Whereas the above definition of an injury includes drowning (lack of oxygen), hypothermia (lack of heat), strangulation (lack of oxygen), decompression sickness or "the bends" (excess nitrogen compounds) and poisonings (by toxic substances), it does NOT include conditions that result from continual stress, such as carpal tunnel syndrome, chronic back pain and poisoning due to infections. Mental disorders and chronic disability, although these may be eventual consequences of physical injury, are also excluded by the above definition."

Although included in the WHO definition, poisonings will be excluded from the CTR as these have been extremely rare events in the CTR to date and are not typically included in trauma registries in most other contexts.

Patients who are not formally admitted and discharged within 24 hours from the Emergency Ward will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A prospective cohort study of all eligible admitted trauma patients in the Cameroon Trauma registry (CTR) and a qualitative study of 110 in-depth interviews (IDIs).
  The 10 study sites of the CTR are as follows:
  1. Laquintinie Hospital of Douala, (Littoral region)
  2. Limbé Regional Hospital, (Southwest region)
  3. Pouma Catholic Hospital, (Littoral region)
  4. Edea Regional Hospital, (Littoral region)
  5. The Emergency and Reanimation Center of Yaounde, (Centre Region)
  6. Bafoussam Regional Hospital (West region)
  7. Maroua Regional Hospital (Far north region)
  8. Bafia district hospital (Centre Region)
  9. Kribi District hospital (South Region)
  10. Bertoua Regional Hospital (East Region)
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of Successful Contacts | 2 weeks post-discharge
  Proportion of hospitalized trauma patients who are reached by mobile phone at 2weeks post-discharge.
Proportion of Successful Contacts | 1 month post-discharge
  Proportion of hospitalized trauma patients who are reached by mobile phone at 1 month post-discharge.
Proportion of Successful Contacts | 3 months post-discharge
  Proportion of hospitalized trauma patients who are reached by mobile phone at 3 months post-discharge.
Proportion of Successful Contacts | 6 months post-discharge
  Proportion of hospitalized trauma patients who are reached by mobile phone at 6 months post-discharge.
Proportion needing follow-up care. | 2 weeks post-discharge
  Proportion of hospitalized trauma patients who are reached by mobile phone at 2 weeks post-discharge and who are identified by the standard screening tool as needing follow-up care.
Proportion needing follow-up care. | 1 month post-discharge
  Proportion of hospitalized trauma patients who are reached by mobile phone at 1 month post-discharge and who are identified by the standard screening tool as needing follow-up care.
Proportion needing follow-up care. | 3 months post-discharge
  Proportion of hospitalized trauma patients who are reached by mobile phone at 3 months post-discharge and who are identified by the standard screening tool as needing follow-up care.
Proportion needing follow-up care. | 6 months post-discharge
  Proportion of hospitalized trauma patients who are reached by mobile phone at 6 months post-discharge and who are identified by the standard screening tool as needing follow-up care.
Proportion needing follow-up care. | 24 months
  Cumulative Proportion of hospitalized trauma patients who are reached by mobile phone over the study period and who are identified by the standard screening tool as needing follow-up care.
Qualitative outcomes: Examine Inner setting of the Consolidated Framework for Implementation Research (CFIR) | 6 months through 24 months
  Examine through qualitative data, the inner setting domain of the Consolidated Framework for Implementation Research (CFIR) among patients, facility staff, and research assistants
Qualitative outcomes: Examine Outer setting of the Consolidated Framework for Implementation Research (CFIR) | 6 months through 24 months
  Examine through qualitative data, the outer setting domain of the Consolidated Framework for Implementation Research (CFIR) among patients, facility staff, and research assistants
Qualitative outcomes: Examine Characteristics of individuals using the Consolidated Framework for Implementation Research (CFIR) | 6 months through 24 months
  Examine through qualitative data, the Characteristics of individuals using the Consolidated Framework for Implementation Research (CFIR) among patients, facility staff, and research assistants
Qualitative outcomes: Examine Process of implementation using the Consolidated Framework for Implementation Research (CFIR) | 6 months through 24 months
  Examine through qualitative data, the process of implementation using the Consolidated Framework for Implementation Research (CFIR) among patients, facility staff, and research assistants.

SECONDARY OUTCOMES:
Disability assessed by Augmented Glasgow Outcomes Scale-Extended (aGOSE) | 24 months; after the last participant recruited in month 18 completes 6 month follow-up.
  Assess disability for the total cohort and subgroups (study site, socioeconomic status, injury mechanism, injury type, participant demographics, hospital type) at each timepoint as determined by Augmented Glasgow Outcomes Scale-Extended (aGOSE). A possible score of 1 through 8; lowest score of 1 means death while maximum score of 8 means Upper good recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Chichom-Mefire, MD, Principal Investigator — University of Buea; Catherine Juillard, MD, MPH, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data for all primary and secondary outcome measures will be made available upon reasonable request to Harnessing Data Science for Health Discovery and Innovation in Africa (DSI Africa) consortium and other researchers.